CLINICAL TRIAL: NCT02581436
Title: Addition of kSORT Assay in the Follow-up of Patients After Kidney Transplantation
Brief Title: Testing Immunosuppression Threshold in Renal Allografts To Extend eGFR
Acronym: TITRATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1217
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Disorder Related to Renal Transplantation; Renal Transplant Rejection; Acute Graft Rejection
Keywords: Prediction test; genetic transcription profile; Transplant follow-up; Chronic index; Graft Function

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- kSORT assay based follow-up (Experimental): Post Transplant surveillance based on the result of the kSORT assay.
  Interventions: Other: kSORT assay based follow-up
- Standard follow-up (Active Comparator): Post Transplant surveillance based on standard of care.
  Interventions: Other: Standard follow-up

INTERVENTIONS:
Other: kSORT assay based follow-up — kSORT assay in pre-established days: 14, 45, 90, 180, 365 and 540 of post transplantation follow-up. If kSORT result is positive maintenance immunosuppressive will be increased (tacrolimus trough levels 12-15 ng/mL, Mofetil Mycophenolate 1.5 mg every 24 hours and prednisone 5 mg/day) and graft biopsy will be obtained. Kidney biopsy will be obtained one mo after treatment as well as kSORT assay. If kSORT result is negative, the maintenance immunosuppressor dosages will remain as established in our institutional guidelines. If after a year of follow-up, the kSORT result is negative, immunosuppression will be decreased (Tacrolimus levels 5 - 10 ng/ml and mofetil mycophenolate 500 mg every 12 hours).
  Arms: kSORT assay based follow-up
Other: Standard follow-up — Surveillance will be the usual, includes creatinine determinations and clinical evaluation as often as established in the institutional protocol. A kidney graft biopsy will be obtained in case of dysfunction (increase in serum creatinine >25% above baseline or 0.3 mg/mL above baseline) or as part of our institutional programmed biopsies (months 3 and 12). Treatment will be established in accordance with biopsy results. In all cases of rejection a kidney biopsy will be obtained one month after initiating treatment. In this control group, samples for kSORT analysis will be collected on pre-established dates for the study, but patient treatment will not be contingent on the assay's results; investigators will be blinded to the result in this control patient group.
  Arms: Standard follow-up

SUMMARY:
This study evaluates the addition of "Kidney Solid Organ Rejection Test" (kSORT), in the clinical follow-up of renal transplant recipients, compared to clinical standard surveillance in the first two years after kidney transplantation. The design of the study is a partially blinded, randomized control trial of patients with living and deceased donor. The recruitment will be in a third level attention hospital in Mexico city (Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán). The main outcomes are the rate and grade of acute rejection, histologic chronic index of the one year protocol biopsy and glomerular filtration rate.

DETAILED DESCRIPTION:
I. Background Kidney transplantation is the treatment of choice in patients with end stage renal disease in need of function replacement therapy, and in whom there is no absolute contraindication to the procedure. The current figures reported in the USA on post-transplant graft survival at one year, are 95% in cases of living donor (LD) recipients and 90% in deceased donor (DD) recipients3; the mean calculated survival of these grafts has increased and is currently 14 years in LD and 11 years in DD recipients. The fact that graft survival hinges on multiple immune and non-immune factors is well recognized; however, the main cause of graft loss is solidly linked to its rejection, with evidence of involvement of the immune humoral response in most cases (specific antibodies against HLA antigens).

The main cause of acute graft dysfunction is acute rejection (AR). Several studies have associated episodes of this entity with chronic structural injury and subsequent functional impairment. Thus, timely diagnostic certainty is pivotal so as to optimize immunosuppressive therapy and preserve graft function. To date, the only tool available to confirm AR is graft biopsy and its established histological diagnostic criteria8. However, this diagnostic tool has limitations resulting mainly from sampling errors and costs. Furthermore, about 10% of patients with normal graft function have evidence of AR in protocol biopsies, so centers that do not use this follow-up modality in kidney transplant recipients (KTR) are unable to document this immune phenomenon. Ideally, an AR non-invasive, diagnostic tool would be of utmost use in KTR follow-up since it would preclude the need for graft biopsies and efficiently support the management of immune suppressors. Therefore, the systematic performance of a highly specific and sensitive assay reflecting AR, would allow for the timely detection of this immune phenomenon compared to the current standard (biopsy). Moreover, the systematic use of a tool with these characteristics would allow stratification of the immunological risk as well as proactive adjustment of immunosuppressor drug dosages, potentially limiting chronic injury and improving the graft's survival.

The background to the proposed study is based on the extensive line of research conducted by Dr. Sarwal et al. They have recently published results10 on monitored pediatric kidney transplant recipients. Biomarkers of gene panels in peripheral blood detected by microarray were discovered in a single institution and subsequently validated by quantitative-PCR in 12 pediatric kidney transplant programs. A total of 367 individual blood samples, each paired to a graft biopsy for blinded centralized classification, were analyzed (115 with acute rejection, 180 with stable kidney graft function, and 72 with other causes of graft injury). Among the genes differentially expressed in microarrays, quantitative-PCR analysis of a set of 5 genes (DUSP1, PBEF1, PSEN1, MAPK9 and NLTR) classified acute rejection with great precision. The 5 gene model has a sensitivity of 91%, specificity of 94%, positive predictive value of 83%, negative predictive value of 97% and a 92% precision when differentiating acute rejection samples from other phenotypes (stable and no acute rejection, no acute rejection/ non-stable). Interestingly, 8/12 samples from patients with borderline rejection on biopsy, were classified as acute rejection with the 5 gene model. The frequent prediction of the phenotype in borderline rejection biopsies suggests that pre-clinical injury in acute rejection could also be identified by quantitative-PCR in peripheral blood samples, thus allowing earlier treatment of these patients.10 The fact that this model predicts acute rejection in both cellular and humoral immune injury modalities, is of utmost relevance. Moreover, these genes in peripheral blood, strongly linked to graft rejection, do not correlate (are independent) with many demographic, clinical, treatment modalities and bacterial/viral infection parameters.

The 5 genes are centered on leukocyte trafficking and T/B cell activation and are mostly expressed in monocytes, activated in the peripheral circulation; they reflect injury response mechanisms to cellular oxidative stress (DUSP1), apoptosis (MAPK9), IL2-dependent cytolytic gene activation (NKTR), increased cell adhesion via the e-cadherin/catenin complex (PSEN1) and smooth muscle vascular cell injury (PBEF1).

The authors pointed out that the study was conducted in a pediatric and young adult population, in whom rejection may be more aggressive due to the disparity between the adult transplanted organ and the pediatric recipient, or as a result of poor treatment adherence in adolescent recipients, leading to a stronger immune response. Thus, the 5-gene model would require further evaluation in order to determine its diagnostic potential of acute rejection in patients of all ages, in larger patient cohorts and in association with different immunosuppressant regimes.

For these reasons, the same group of investigators undertook a large study to identify a transcription profile that would unify the kidney transplant recipient population independently of age, the cause of terminal renal disease, comorbidities, and the type of immune suppression used in different centers in the USA, Mexico and Europe. The final selection of 17 genes included 10 genes in the pediatric population and 7 newly identified genes and allowed the molecular classification of acute rejection in adult and pediatric patients. They correctly predicted the presence of acute rejection and non-acute rejection in the different samples collected from patients in various participating study sites, and in recipients of different ages with no previous data normalization. On the basis of these observations, a score was generated using 14 of the 17 genes, and with Pearson's correlation test, a score was attributed to each detected gene and compared with the genetic profile found in patients with and without rejection, assigning the number +1 or -1. The score ranges between -13 and +13. Among the patients in whom the score predicted a "high risk of rejection" (Acute Rejection Risk-Score ≥ 7), 90.24% were correctly classified as acute rejection, while if the test predicted "a very low risk of acute rejection" (Acute Rejection Risk-Score ≤ -7), 97.7% were correctly classified as non-acute rejection on the basis of the biopsy findings. Furthermore, the average predictive probability of acute rejection was highly significant when comparing acute rejection vs. non-acute rejection in 4 centers (p<0.0001; p=0.002; p<0.0001; p<00001), respectively. This model equally detected acute rejections mediated by antibodies as well as those that were cell-mediated, with a high predictive probability. The prediction of acute rejection was independent of the post-transplant period duration. These 17 genes are included in the KSORT assay (Kidney Solid Organ Rejection Test) and the algorithm generating the risk score is known as the kSORT analysis suit (kSAS).

In a recently published study with data from our Institute, in which the results of biopsies obtained because of post-transplant dysfunction were reviewed between January 2007 and December 2011 (n=223), we observed an AR incidence during the first year post-transplant of 11.8% in live donor KTR and of 17.4% in deceased donor graft recipients. Throughout 2013, the number of kidney transplants performed at the Institute increased to 63 (53% from living donors, 46% from deceased donors). In accordance with our institutional protocol for the follow-up of kidney transplant recipients, we currently obtain protocol graft biopsies on the 3rd and 12th month post-transplant. The protocol biopsies are obtained at established timepoints with the purpose of documenting whether there is any evidence of immunological activity (sub-clinical) or signs of other pathologies that would require modification of the immunosuppressive therapeutic regime. We also obtain a graft biopsy at any point in the post-transplant period if abnormalities in renal function develop, defined as a verified increase in serum creatinine ≥ 25% over previous baseline values, and in the absence of other evident pathologies such as obstructive processes of the urinary tract, urinary tract infections, dehydration, supra-therapeutic blood levels of the used calcineurin inhibitor.

As of May 2013, the date in which the 3rd month protocol biopsy was established, we have documented an incidence of sub-clinical acute rejections, including borderline and major rejections according to the Banff classification, of 52% (10/40 biopsies revealed acute cellular or humoral rejection and 11/40 had borderline injury). This number is unprecedented at the Institute because protocol biopsies were not previously obtained on the 3rd month.

Currently, all KTR at the Institute receive an induction therapy modality (Thymoglobulin or Basiliximab), depending on their individual immunological risk and the origin of the graft. Hence, all live donor KT recipients with a PRA <30% and no HLA donor specific antibodies (DSA) are treated with Basiliximab (anti-IL2R monoclonal antibody; 2 doses of 20mg each); the exceptions are KTR sharing 2 haplotypes with their donor and that receive no induction therapy. All deceased donor graft recipients (independently of the PRA %), live donor KTR with positive donor-specific HLA antibodies (independently of the PRA %) or with a PRA ≥30%, are induced with Thymoglobulin (rabbit polyclonal antibody preparation, at a total dose of 4.5mg/Kg). All patients must have a lymphocyte crossmatch test (T/B), a negative CDC-AHG and those with DSA (Single antigen, Luminex) also require a negative crossmatch by flow cytometry.

Biopsy-proven acute rejection events are treated with pulses of methylprednisolone for 3 consecutive days. Patients with steroid-resistant acute cellular rejection (biopsy-proven), are administered Thymoglobulin (1.5 mg/Kg/body weight, for 7 days). Patients with antibody-mediated acute rejection (humoral rejection) are treated with 3-5 plasmapheresis (PP) sessions, 100 mg IV Ig per Kg body weight after each PP session and rituximab (anti-CD20 monoclonal antibody) at the end of all PP sessions.

The standard initial and maintenance immunosuppressive regime is Tacrolimus, Mofetil Mycophenolate and prednisone. The initial Tacrolimus doses are aimed to obtain blood trough levels of 10 to 15 ng/mL, until the 3rd month post-transplant; subsequently and in the absence of AR during the first trimester (clinical or by protocol biopsy), the trough levels are maintained between 8 and 10 ng/mL throughout the first year post-transplant. The maintenance dose of prednisone is 5 mg daily and that of Mofetil Mycophenolate is 1-1.5 g daily.

II. Justification In previous paragraphs, we described the KSORT test's high sensitivity and specificity in the detection of acute rejection. It is now necessary to attempt its transfer into the clinical setting and to help support treatment decisions, such as increasing immune suppression based on a positive test result. The impact of this maneuver on efficacy and safety outcomes will be pivotal in order to incorporate this scrutinizing method into daily clinical practice. Our Institute has transplanted over 60 patients in the last few years, so conducting this study in our center is feasible.

III. Hypothesis and aims Hypothesis Adding the kSORT genetic panel to the post-transplant follow-up will decrease the incidence and severity of acute rejection as well as the chronicity indices in the yearly protocol biopsy, and will improve the calculated glomerular filtration rate after a follow-up of two years.

Aims:

To evaluate the safety and efficacy of adding the kSORT test to the surveillance of patients after kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant recipients from living or deceased donor from National Institute of Health and Nutrition Salvador Zubirán

Exclusion Criteria:

* Kidney transplant recipients who have contraindication to graft biopsy. (coagulopathy, anticoagulant therapy or double antiaggregation)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence and grade of biopsy-proven acute rejection | two years
  Based in BANFF 2013 classification, of allograft biopsies obtained during the study period
Chronic index in one year protocol biopsy | One year
  interstitial fibrosis, tubular atrophy and chronic histomorphometry parameters
Calculated glomerular filtration rate | One and two years
  Calculated glomerular filtration rate with MDRD-IDMS formula

SECONDARY OUTCOMES:
Describe the behavior of the assay throughout the follow-up period. | Two years
  Describe the behavior of kSORT assay, risk factors and consequences
Determine the impact of time with positive or negative kSORT assays on the main outcomes | two years
  Determine the impact of time with positive or negative kSORT assays on the main outcomes
Describe the behavior of the assay after the maneuver of increasing or tapering immunosuppression and after treatment of acute rejection. | Two years
Establish the sensitivity and specificity of the kSORT assay in the detection of acute rejection | Two years
Analyze gene expression relating to renal tissue inflammation and fibrosis at the time of the one-year protocol biopsy, and their relation to clinical variables including the previous and current kSORT assay results. | One year
Hospitalization Rate | Two years
  Rate of hospitalization and causes
Viral Infection rate | Two years
  BK virus nephritis, cytomegalovirus infection, adenovirus and herpes zoster.
Graft loss rate | two years
  Graft loss rate, causes,including patient deaths.

OTHER OUTCOMES:
Immunosuppression dosage, levels and brands | Two years
  Establish the assay's impact on the tacrolimus trough levels main outcome as well as on the specific brand, including the number of brand changes. We will correlate the doses and brands, and the number of brand changes of mofetil mycophenolate.
Population genetics | Two years
  Impact on the main outcomes of the population genetics, measured as major histocompatibility complex alleles and haplotipes.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Medical Sciences and Health Salvador Zubiran, Mexico City, D.F., Mexico

IPD SHARING:
Plan to Share IPD: No
At this moment there is no plan to make individual participant data available

REFERENCES:
- [Background] Thierry A, Thervet E, Vuiblet V, Goujon JM, Machet MC, Noel LH, Rioux-Leclercq N, Comoz F, Cordonnier C, Francois A, Marcellin L, Girardot-Seguin S, Touchard G. Long-term impact of subclinical inflammation diagnosed by protocol biopsy one year after renal transplantation. Am J Transplant. 2011 Oct;11(10):2153-61. doi: 10.1111/j.1600-6143.2011.03695.x. Epub 2011 Aug 22. PMID 21883902
- [Result] Sellares J, de Freitas DG, Mengel M, Reeve J, Einecke G, Sis B, Hidalgo LG, Famulski K, Matas A, Halloran PF. Understanding the causes of kidney transplant failure: the dominant role of antibody-mediated rejection and nonadherence. Am J Transplant. 2012 Feb;12(2):388-99. doi: 10.1111/j.1600-6143.2011.03840.x. Epub 2011 Nov 14. PMID 22081892
- [Result] Meier-Kriesche HU, Ojo AO, Hanson JA, Cibrik DM, Punch JD, Leichtman AB, Kaplan B. Increased impact of acute rejection on chronic allograft failure in recent era. Transplantation. 2000 Oct 15;70(7):1098-100. doi: 10.1097/00007890-200010150-00018. PMID 11045649
- [Result] Pallardo Mateu LM, Sancho Calabuig A, Capdevila Plaza L, Franco Esteve A. Acute rejection and late renal transplant failure: risk factors and prognosis. Nephrol Dial Transplant. 2004 Jun;19 Suppl 3:iii38-42. doi: 10.1093/ndt/gfh1013. PMID 15192134
- [Result] Li L, Khatri P, Sigdel TK, Tran T, Ying L, Vitalone MJ, Chen A, Hsieh S, Dai H, Zhang M, Naesens M, Zarkhin V, Sansanwal P, Chen R, Mindrinos M, Xiao W, Benfield M, Ettenger RB, Dharnidharka V, Mathias R, Portale A, McDonald R, Harmon W, Kershaw D, Vehaskari VM, Kamil E, Baluarte HJ, Warady B, Davis R, Butte AJ, Salvatierra O, Sarwal MM. A peripheral blood diagnostic test for acute rejection in renal transplantation. Am J Transplant. 2012 Oct;12(10):2710-8. doi: 10.1111/j.1600-6143.2012.04253.x. PMID 23009139
- [Result] Roedder S, Sigdel T, Salomonis N, Hsieh S, Dai H, Bestard O, Metes D, Zeevi A, Gritsch A, Cheeseman J, Macedo C, Peddy R, Medeiros M, Vincenti F, Asher N, Salvatierra O, Shapiro R, Kirk A, Reed EF, Sarwal MM. The kSORT assay to detect renal transplant patients at high risk for acute rejection: results of the multicenter AART study. PLoS Med. 2014 Nov 11;11(11):e1001759. doi: 10.1371/journal.pmed.1001759. eCollection 2014 Nov. PMID 25386950